CLINICAL TRIAL: NCT04281706
Title: Impact of Etomidate vs. Propofol on Development of Sepsis and Infectious Complications Post Cardiac Surgery
Brief Title: Impact of Etomidate vs. Propofol on Infectious Complications Post Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Felix Balzer, Prof. Dr. Dr. Felix Balzer, MSc; ECDF-Professor for, Charite University, Berlin, Germany
Other Study IDs: EtoProp
Record Dates: First submitted 2020-01-27; First posted 2020-02-24 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Etomidate-Time-Frame: Patients that underwent cardiac surgery between October 1st, 2012 and September 30th, 2013
  Interventions: Drug: Etomidate vs Propofol as induction agent
- Propofol-Time-Frame: Patients that underwent cardiac surgery between February 1st, 2014 and January 31st, 2015
  Interventions: Drug: Etomidate vs Propofol as induction agent

INTERVENTIONS:
Drug: Etomidate vs Propofol as induction agent — Patients undergoing cardiac surgery were induced with Etomidate according to the standard operating procedure for induction until October 1st, 2013, afterwards a new SOP with Propofol as primary induction agent was introduced. After a washout period of 3 months, Propofol was used as sole induction agent. The rest of the standard operating procedure remained the same.

SUMMARY:
The aim of this retrospective before-after-study is to evaluate the potential association of etomidate vs. propofol as an induction agent for major cardiac surgery on infectious post-operative complications.

The investigators hypothesize that etomidate increases the rate post-operative infectious complications in cardiosurgical patients.

DETAILED DESCRIPTION:
Etomidate had been a standard induction agent as it results in increased hemodynamic stability compared to propofol. This is seen as a major advantage in patients that frequently have a fragile haemodynamic situation.

A major side effect of Etomidate is the resulting adrenal dysfunction, which hampers the bodies stress response and has been shown to cause a higher mortality in infectious contexts such as sepsis. It remains unclear to what extend this attenuated stress response has an impact on the post-operative context in cardiosurgical patients. First preliminary data show that patients receiving Etomidate as an induction agent are more prone to infection than those receiving a different agent, a definitive correlation is nevertheless still lacking.

This is a retrospective before-after-study comparing the rate of infectious complications in patients receiving either valve and/or coronary cardiac surgery at the Charité - Universitätsmedizin Berlin between October 1st, 2012 and January 31th, 2015. On October 1st, 2013 the standard operating procedures for anesthesia for cardiac surgery were amended and the induction agent at the Charité - Universitätsmedizin Berlin was switched from Etomidate to Propofol. The investigators are therefore comparing patients undergoing cardiac surgery between October 1st, 2012 and September 30th, 2013 as the Etomidate group with patients undergoing surgery between February 1st, 2014 and January 31st, 2015 as the Propofol group. The gap in between the two groups (October 1st, 2013 - January 31st, 2014) was defined as a washout phase to account for a potential delay in implementation of the renewed standard operating procedures. Patients will be investigated unmatched as well as matched according to (Age, Body Mass Index, American Society of Anesthesiologists physical status classification system (ASA), New York Heart Association Functional Classification (NYHA), Surgical Mode and Diabetes). The data for both groups will be acquired from the 2 electronic patient data management systems at our hospital (COPRA System, Sasbachwalden, Germany, and SAP, Walldorf, Germany).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Valve and/or coronary artery bypass graft surgery

Exclusion Criteria:

* Surgery during washout period (October 1st, 2013 - January 31st, 2014)
* Resurgery
* Endocarditis
* Known immunosuppression:
* Corticosteroid therapy
* Solid organ transplant
* Stem Cell therapy
* HIV diagnosis

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — all gender are eligible.
Study Population: Patients that underwent cardiac surgery between October 1st, 2012 and January 31st, 2015
Sampling Method: Non-Probability Sample
Enrollment: 1495 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Sepsis | surgical intervention to hospital discharge, average 30 days
  Incidence of sepsis according to diagnosis-related group coding between surgical intervention and hospital discharge (according to SEPSIS II)

SECONDARY OUTCOMES:
Pneumonia | surgical intervention to hospital discharge, average 30 days
  Incidence of pneumonia within between surgical intervention and hospital discharge
Mediastinitis | surgical intervention to hospital discharge, average 30 days
  Incidence of mediastinitis within between surgical intervention and hospital discharge
Surgical Site Infections | surgical intervention to hospital discharge, average 30 days
  Incidence of surgical site infections between surgical intervention and hospital discharge
ICU Mortality | surgical intervention to ICU discharge, average 30 days
  Proportion of patients that died before ICU discharge
Hospital mortality | surgical intervention to hospital discharge, average 30 days
  Proportion of patients that died before hospital discharge
Intensive Care Unit length of stay | ICU admission to ICU discharge, average 30 days
  Time patients spend on the ICU
Hospital length of stay | hospital admission to hospital discharge, average 30 days
  Time patients spend admitted to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Dr. Felix Balzer, MSc, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité - Universitätsmedizin Berlin, Corporate Member of Freie Universität Berlin, Humboldt Universität zu Berlin and Berlin Institute of Health, Augustenburger Platz 1, 13353, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No